CLINICAL TRIAL: NCT05762744
Title: Pharmacogenomics of GLP1 Receptor Agonists
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We concluded that it would not be possible to meet our recruitment targets within the available budget. The study was ended when the funding ended.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Simeon I. Taylor, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HP-00067574
Record Dates: First submitted 2023-02-23; First posted 2023-03-10 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: GLP1; insulin; glucose; exenatide; GLP1 receptor agonist; insulin secretion; glucagon receptor; GIP receptor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Exenatide

STUDY DESIGN:
Intervention Model Description: Research participants all received the same two interventions (saline or exenatide) but the order of the interventions was randomized.
Who Masked: Participant
Masking Description: Participants were not informed whether the nurse was administering saline or exenatide injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exenatide followed by saline (Other): Participants were randomized to receive exenatide 15 min before the first frequently sampled iv glucose tolerance test and saline 15 min before the second frequently sampled iv glucose tolerance test
  Interventions: Drug: Exenatide Injection (before the first FSIGT)
- Saline followed by exenatide (Other): Participants were randomized to receive saline15 min before the first frequently sampled iv glucose tolerance test and exenatide15 min before the second frequently sampled iv glucose tolerance test
  Interventions: Drug: Exenatide injection before the second FSIGT)

INTERVENTIONS:
Drug: Exenatide Injection (before the first FSIGT) — Nurses administered exenatide (5 mcg) subcutaneously 15 minutes prior to conducting the first frequently sampled intravenous glucose tolerance test.
  In this crossover study, participants will also be "crossed over" to receive saline rather than exenatide: Nurses administered saline (0.2 mL) subcutaneously 15 minutes prior to conducting a frequently sampled intravenous glucose tolerance test.
  Other Names: BYETTA; Exenatide
  Arms: Exenatide followed by saline
Drug: Exenatide injection before the second FSIGT) — Nurses administered exenatide (5 mcg) subcutaneously 15 minutes prior to conducting the second frequently sampled intravenous glucose tolerance test.
  Other Names: BYETTA; Exenatide
  Arms: Saline followed by exenatide

SUMMARY:
Healthy volunteers were recruited from the Old Order Amish population in Lancaster County, Pennsylvania. After providing informed consent, research participants were screened for eligibility. The clinical trial was designed as a randomized crossover study in which participants underwent two frequently sampled intravenous glucose tolerance tests - one after receiving a subcutaneous injection of saline and one after receiving a subcutaneous injection of rapid-acting exenatide (BYETTA). The study sought to determine whether genetic variants are associated with the magnitude of the effect of exenatide. However, because the study fell far short of its recruitment targets, it was under-powered to evaluate genetic association. Thus, the data analysis focused on testing the hypothesis that the order of testing (whether the placebo FSIGT was conducted before the exenatide-stimulated FSIGT or whether the FSIGTs were conducted in the reverse order) does not alter the magnitude impact of exenatide on responses to a frequently sampled iv glucose tolerance test.

DETAILED DESCRIPTION:
Healthy volunteers were recruited from the Old Order Amish population in Lancaster County, Pennsylvania. After providing informed consent, research participants were screened for eligibility. The clinical trial was designed as a randomized crossover study in which participants underwent two frequently sampled intravenous glucose tolerance tests (FSIGT) - one after receiving a subcutaneous injection of saline and one after receiving a subcutaneous injection of rapid-acting exenatide (BYETTA). Based on data obtained from the FSIGT, participants' response to exenatide was assessed -- specifically, the effect of exenatide to enhance insulin secretion and accelerate metabolism of glucose. The study sought to determine whether genetic variants are associated with the magnitude of the effect of exenatide. However, because the study fell far short of its recruitment targets, it was under-powered to evaluate genetic association. Thus, the data analysis focused on testing the hypothesis that the order of testing (whether the placebo FSIGT was conducted before the exenatide-stimulated FSIGT or whether the FSIGTs were conducted in the reverse order) does not alter the magnitude impact of exenatide on responses to a frequently sampled iv glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Old Order Amish community in Lancaster County, Pennsylvania
* BMI: 18-40 kg/sq.m.

Exclusion Criteria:

* Known allergy to exenatide
* History of diabetes, random glucose >200 mg/dL, or HbA1c > 6.5%
* Significant debilitating chronic cardiac, hepatic, pulmonary, or renal disease or other diseases that the investigator judges will make interpretation of the results difficult or increase the risk of participation
* Seizure disorder
* Pregnant by self-report or known pregnancy within 3 months of the start of study
* Currently breast feeding or breast feeding within 3 months of the start of the study
* Estimated glomerular filtration rate <60 mL/min/1.73m2
* Hematocrit <35%
* Liver function tests greater than 2 times the upper limit of normal
* Abnormal thyroid stimulating hormone
* History of pancreatitis or pancreatic cancer. Personal or family history of medullary carcinoma of the thyroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 63 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simeon I Taylor, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Amish Research Clinic, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Subject to protection of confidential information of research participants, we will share data with qualified researchers.
Supporting Information: ICF
Time Frame: 12 months after publication in a peer reviewed journal.
Access Criteria: Must sign data transfer agreement to protect confidentiality of research participants.
  Requester must be on faculty at an accredited academic institution such as a medical school.

REFERENCES:
- [Background] Taylor SI, Montasser ME, Yuen AH, Fan H, Yazdi ZS, Whitlatch HB, Mitchell BD, Shuldiner AR, Muniyappa R, Streeten EA, Beitelshees AL. Acute pharmacodynamic responses to exenatide: Drug-induced increases in insulin secretion and glucose effectiveness. Diabetes Obes Metab. 2023 Sep;25(9):2586-2594. doi: 10.1111/dom.15143. Epub 2023 Jun 1. PMID 37264484
- [Derived] Beitelshees AL, Streeten EA, Shahidzadeh Yazdi Z, Whitlatch HB, Mitchell BD, Shuldiner AR, Montasser ME, Taylor SI. Acute pharmacodynamic responses to sitagliptin: Drug-induced increase in early insulin secretion in oral glucose tolerance test. Clin Transl Sci. 2024 May;17(5):e13809. doi: 10.1111/cts.13809. PMID 38700326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates: June 2016 - November 2018 Site: Community-based recruitment at Amish Research Clinic, Lancaster Pennsylvania (Univ. of Maryland School of Medicine)
Pre-assignment Details: Participants were assigned to specific arms of the study based on the order in which they were randomized to a subcutaneous injection of either exenatide or normal saline solution:
  Arm 1: Exenatide followed by Normal Saline Arm 2: Normal Saline followed by Exenatide Frequently sampled intravenous glucose tolerance tests (FSIGT) were initiated 15 minutes after the subcutaneous injections of exenatide or normal saline. The second FSIGT was performed 5-28 days after the first FSIGT.
Groups:
- Exenatide Followed by Normal Saline: Of the 54 participants in our study, 26 individuals were randomized to receive exenatide 15 min before the first frequently sampled intravenous glucose tolerance test (FSIGT) and saline 15 min before the second FSIGT
- Normal Saline Followed by Exenatide: Of the 54 participants in our study, 26 individuals were randomized to receive normal saline 15 min before the first frequently sampled intravenous glucose tolerance test (FSIGT) and exenatide 15 min before the second FSIGT
Period: 1st iv Glucose Tolerance Test
Arm/Group | Exenatide Followed by Normal Saline | Normal Saline Followed by Exenatide
Started | 31 | 32
Completed | 26 | 26
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Some critical blood samples not collecte | 5 | 5
Period: 2nd iv Glucose Tolerance Test
Arm/Group | Exenatide Followed by Normal Saline | Normal Saline Followed by Exenatide
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Because the primary outcomes focused on the effects of exenatide, we restricted the analysis to participants who completed both periods of the study (i.e., both the exenatide-stimulated and the comparator placebo studies).
Groups:
- Exenatide First Followed by Normal Saline: Exenatide (5 mcg, sc) was injected 15 minutes before the first frequently sampled iv glucose tolerance test (FSIGT). After a washout period of 5-28 days, participants underwent a second FSIGT with saline (0.20 mL) being injected 15 min before the 2nd FSIGT.
- Normal Saline Followed by Exenatide: Saline (0.2 mL) was injected 15 minutes before the first frequently sampled iv glucose tolerance test (FSIGT). After a washout period of 5-28 days, participants underwent a second FSIGT with exenatide (5 mcg) being injected 15 min before the 2nd FSIGT.
- Total: Total of all reporting groups
Arm/Group | Exenatide First Followed by Normal Saline | Normal Saline Followed by Exenatide | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Full Range); unit: Years] | 50.2 [24 to 72] | 44.6 [28 to 66] | 47.3 [24 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 18 | 13 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 26 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (3.8) | 27.8 (3.7) | 28.1 (3.7)
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of glycated hemoglobin] | 5.6 (0.4) | 5.5 (0.3) | 5.5 (0.3)
Number of participants homozygous for major alleles of both GCGR and GIPR [Count of Participants; unit: Participants] | 9 | 10 | 19
Number of participants homozygous for p.G40S allele of GCGR [Count of Participants; unit: Participants] | 12 | 8 | 20
Number of participants homozygous for p.E354Q allele of GIPR [Count of Participants; unit: Participants] | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Exenatide Effect on First Phase Insulin Secretion
Description: The ratio of the area-under-the-curve (AUC) for 1st phase insulin secretion in the exenatide-stimulated FSIGT divided by the AUC for 1st phase insulin secretion in the saline FSIGT.
Time Frame: 0-10 minutes
Population: The analysis population included 52 patients who completed the study and for whom the necessary blood samples were collected and available for assays of insulin and glucose.
Measure: Mean (Standard Error); unit: Ratio (no units)
Groups:
- Exenatide First Followed by Saline: Participants who were randomized to undergo exenatide-stimulated FSIGT first followed by saline FSIGT
- Saline First Followed by Exenatide: Participants who were randomized to undergo the saline FSIGT followed by the exenatide-stimulated FSIGT
Arm/Group | Exenatide First Followed by Saline | Saline First Followed by Exenatide
Number analyzed (Participants) | 26 | 26
Ratio (no units) | 1.90 (0.17) | 2.18 (0.25)
Statistical Analysis 1: Comparison: Exenatide First Followed by Saline vs Saline First Followed by Exenatide; Null hypothesis: the order of FSIGTs (saline or exenatide-stimulated) does not affect the response during an FSIGT; Test type: Other — Unpaired two-tailed t-test to test null hypothesis; p = 0.37, t-test, 2 sided — The t-test was conducted on the logarithms of the variable

2. Primary Outcome: Exenatide Effect on Glucose Disappearance Rate
Description: The ratio of the glucose disappearance rate (exenatide) divided by the glucose disappearance rate (placebo).
  Glucose disappearance rates were calculated as the slope of the plot of the logarithm of the glucose concentration as a function of time.
Time Frame: 25-50 minutes
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Ratio (no units)
Groups:
- Exenatide First Followed by Saline: Participants who were randomized to undergo the exenatide-stimulated FSIGT first followed by saline FSIGT
- Saline First Followed by Exenatide: Participants who were randomized to undergo the saline FSIGT first followed by the exenatide-stimulated FSIGT
Arm/Group | Exenatide First Followed by Saline | Saline First Followed by Exenatide
Number analyzed (Participants) | 26 | 26
Ratio (no units) | 2.16 (0.19) | 2.28 (0.20)
Statistical Analysis 1: Comparison: Exenatide First Followed by Saline; Null hypothesis: The order of FSIGT (exenatide-stimulated or saline) does not affect the response to an FSIGT; Test type: Other — Two-tailed unpaired t-test to test null hypothesis; p = 0.66, t-test, 2 sided

3. Secondary Outcome: Glucose Disappearance Rate (Exenatide)
Description: The slope of the line plotting the logarithm of glucose concentrations as a function of time during the exenatide frequently sampled intravenous glucose tolerance test. The slope of the line was estimated as the slope of the least-squares fit to the data points between 25-50 minutes.
Time Frame: 25-50 minutes
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log(mg/dL) per min
Groups:
- Exenatide First Followed by Saline: Participants who were randomized to undergo exenatide-stimulated FSIGT first followed by a saline FSIGT
- Saline First Followed by Exenatide: Participants who were randomized to undergo a saline FSIGT first followed by an exenatide-stimulated FSIGT
Arm/Group | Exenatide First Followed by Saline | Saline First Followed by Exenatide
Number analyzed (Participants) | 26 | 26
Log(mg/dL) per min | 1056 (94) | 1131 (81)
Statistical Analysis 1: Comparison: Exenatide First Followed by Saline vs Saline First Followed by Exenatide; Null hypothesis: the order of testing (exenatide-stimulated or saline FSIGT) does not affect data obtained in the FSIGTs; Test type: Other — Two-tailed unpaired t-test to test null hypothesis; p = 0.55, t-test, 2 sided

4. Secondary Outcome: Glucose Disappearance Rate (Placebo)
Description: The slope of the line plotting the logarithm of glucose concentrations as a function of time during the placebo frequently sampled intravenous glucose tolerance test. The slope of the line was estimated as the slope of the least-squares fit to the data points between 25-50 minutes.
Time Frame: 25-50 minutes
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Log(mg/dL) per min
Groups:
- Exenatide First Followed by Saline: Participants randomized to undergo the exenatide-stimulated FSIGT first followed by the saline FSIGT.
Arm/Group | Exenatide First Followed by Saline | Saline First Followed by Exenatide
Number analyzed (Participants) | 26 | 26
Log(mg/dL) per min | 500 (37) | 547 (48)
Statistical Analysis 1: Comparison: Exenatide First Followed by Saline vs Saline First Followed by Exenatide; The order of FSIGTs (exenatide-stimulated or saline) does not affect the response during an FSIGT; Test type: Other — Unpaired, two-tailed t-test to test the null hypothesis; p = 0.45, t-test, 2 sided

5. Secondary Outcome: First Phase Insulin Secretion (Exenatide)
Description: The area under the curve for plasma insulin levels during a frequently sampled intravenous glucose tolerance test after participants received exenatide
Time Frame: 0-10 minutes
Population: as for outcome 1
Measure: Mean (Standard Error); unit: microunits/mL*min
Groups:
- Exenatide First Followed by Saline: Participants who were randomized to undergo the exenatide-stimulated FSIGT first followed by the saline FSIGT
- Saline Followed by Exenatide: Participants who were randomized to undergo the saline FSIGT first followed by the exenatide-stimulated FSIGT
Arm/Group | Exenatide First Followed by Saline | Saline Followed by Exenatide
Number analyzed (Participants) | 26 | 26
microunits/mL*min | 561 (94) | 494 (50)
Statistical Analysis 1: Comparison: Exenatide First Followed by Saline vs Saline Followed by Exenatide; Null hypothesis: the order of FSIGT (exenatide or saline) does not affect the response during an FSIGT; Test type: Other — Two-tailed unpaired t-test to test null hypothesis; p = 0.86, t-test, 2 sided — The t-test was conducted on the logarithms of the variable

6. Secondary Outcome: First Phase Insulin Secretion (Placebo)
Description: The area under the curve for plasma insulin levels during a frequently sampled intravenous glucose tolerance test after participants received saline
Time Frame: 0-10 minutes
Population: as for outcome 1
Measure: Mean (Standard Error); unit: microunits/mL*min
Groups:
- Exenatide First Followed by Normal Saline: This includes participants who were randomized to undergo the exenatide-stimulated FSIGT followed by the placebo FSIGT.
- Placebo First Followed by Exenatide: This includes participants who were randomized to receive the placebo FSIGT first followed by the exenatide-stimulated FSIGT
Arm/Group | Exenatide First Followed by Normal Saline | Placebo First Followed by Exenatide
Number analyzed (Participants) | 26 | 26
microunits/mL*min | 305 (38) | 254 (23)
Statistical Analysis 1: Comparison: Exenatide First Followed by Normal Saline vs Placebo First Followed by Exenatide; Null hypothesis: The order of FSIGTs (exenatide-stimulated or saline) does not affect the response to an FSIGT; Test type: Other — Two-tailed p-test for unpaired data; p = 0.44, t-test, 2 sided — The t-test was conducted on the logarithms of the variable

7. Secondary Outcome: Drug Effect on First-Phase Insulin Secretion (Genotype-specific)
Description: The effect of exenatide to increase first-phase insulin secretion was defined as the ratio of area-under-the-curve (AUC) for insulin levels during the first 10 minutes of the exenatide-stimulated FSIGT divided by the AUC for first phase insulin secretion during the saline FSIGT..
Time Frame: 0 - 10 min during the FSIGT
Population: Participants with the specified genotypes. Based on the observation that the order of FSIGT (exenatide-first versus saline-first) did not affect the data obtained in the FSIGT, we have pooled data from the two arms of the study (exenatide-first and saline-first).
Measure: Mean (Standard Error); unit: Ratio: no units
Groups:
- Major Allele Homozygotes: Participant who are homozygous for the major alleles of both GCGR and GIPR. Based on the observation that the order of the two FSIGTs was not associated with significant differences in data from the FSIGT, we pooled data from both arms of the study (exenatide first and saline first).
- Homozygotes for the p.G40S Allele of GCGR: Participants with two copies of the p.G40S allele of GCGR
- Homozygotes for the p.E354Q Allele of GIPR: Participants with two copies of the p.E354Q allele of the GIPR gene
Arm/Group | Major Allele Homozygotes | Homozygotes for the p.G40S Allele of GCGR | Homozygotes for the p.E354Q Allele of GIPR
Number analyzed (Participants) | 19 | 20 | 13
Ratio: no units | 2.25 (0.31) | 1.94 (0.21) | 1.87 (0.27)
Statistical Analysis 1: Comparison: Major Allele Homozygotes vs Homozygotes for the p.G40S Allele of GCGR; Null hypothesis: no differences between the two groups with respect to exenatide's effect on first-phase insulin secretion. t-test conducted on logarithms of the values; Test type: Other; p = 0.41, t-test, 2 sided
Statistical Analysis 2: Comparison: Major Allele Homozygotes vs Homozygotes for the p.E354Q Allele of GIPR; Null hypothesis: no difference between two groups with respect to exenatide's effect on first phase insulin secretion; Test type: Other; p = 0.38, t-test, 2 sided

8. Secondary Outcome: Exenatide's Effect on the Rate of Glucose-disappearance (Genotype Specific)
Description: The rate of glucose disappearance was calculated as the slope of a least-squared line fitted to the logarithms of glucose concentrations during time 25-50 min of FSIGTs
Time Frame: 25-50 min during the FSIGT
Population: Same as for effect of exenatide on first phase insulin secretion
Measure: Mean (Standard Error); unit: Log(mg/dL) per min
Arm/Group | Major Allele Homozygotes | Homozygotes for the p.G40S Allele of GCGR | Homozygotes for the p.E354Q Allele of GIPR
Number analyzed (Participants) | 19 | 20 | 13
Log(mg/dL) per min | 2.19 (0.24) | 2.28 (0.24) | 2.18 (0.19)
Statistical Analysis 1: Comparison: Major Allele Homozygotes vs Homozygotes for the p.G40S Allele of GCGR; Null hypothesis: the two genotype groups do not differ with respect to the effect of exenatide on the rate of glucose disappearance; Test type: Other; p = 0.80, t-test, 2 sided
Statistical Analysis 2: Comparison: Major Allele Homozygotes vs Homozygotes for the p.E354Q Allele of GIPR; Null hypothesis: the two genotype groups do not differ with respect to the effect of exenatide on the rate of glucose disappearance during an FSIGT; Test type: Other; p = 0.98, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the time (one day) participants were in the clinic for the frequently sampled intravenous glucose tolerance test
Description: Participants were interviewed by nursing staff on the day of the frequently sampled intravenous glucose tolerance test.
Groups:
- Total Study Population (Control Study): The analysis is based on observations during the control studies in the 62 individuals who completed the control intravenous glucose tolerance testing. We report the adverse events separately for the control studies versus the exenatide studies because the literature documents the fact that GLP1R agonists like exenatide frequently induce nausea and/or vomiting.
- Total Study Population (Exenatide Study): The analysis is based on observations during the control studies in the 62 individuals who completed exenatide intravenous glucose tolerance testing. We report the adverse events separately for the control studies versus the exenatide studies because the literature documents the fact that GLP1R agonists like exenatide frequently induce nausea and/or vomiting.
Arm/Group | Total Study Population (Control Study) | Total Study Population (Exenatide Study)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 3/62 | 7/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Study Population (Control Study) (N=62) | Total Study Population (Exenatide Study) (N=62)
Nausea or vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) — Participants were interviewed while they were in the clinic undergoing frequently sampled intravenous glucose tolerance test.
Headache (Vascular disorders) | 2 (2) | 4 (4) — Participants were interviewed by nursing staff while participants were in Clinic undergoing frequently sampled intravenous glucose tolerance test.

LIMITATIONS AND CAVEATS:
The study was terminated before achieving the recruitment targets of 24 participants for each genotype group. Thus, the study was under-powered. The data analysis tested the null hypothesis that the order in which participants received exenatide or normal saline does not affect the response to a frequently sampled intravenous glucose tolerance test.

The database is too small to permit meaningful analysis of the incidence of relatively minor adverse events (headaches, nausea, and vomiting).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT05762744/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT05762744/ICF_001.pdf